CLINICAL TRIAL: NCT04506437
Title: Foster Care Mental Health Family Navigator
Acronym: FCFN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R34MH119433-01A1 (NIH); 1R34MH119433-01A1 (NIH)
Record Dates: First submitted 2020-08-06; First posted 2020-08-10 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Mental Health
Keywords: Adolescent; Foster Care; Mental Health; Navigator; Service Access
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: This is a dynamic wait-listed design in which the investigators will test a theory-driven family-based navigator treatment engagement intervention (FCFN) while also collecting data on the FCFN model's potential implementation and adoption within child welfare and behavioral health settings.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Family-based mental health navigation (Experimental): Family-based navigator intervention combined with mHealth practices to improve mental health treatment initiation and engagement
  Interventions: Behavioral: Family-based mental health navigation
- Standard of care, then family-based mental health navigation (Active Comparator): During wait-list period receive standard of care engagement practices and services-as-usual, and after the wait-list period the participants receive the family-based navigator intervention combined with mHealth practices
  Interventions: Behavioral: Family-based mental health navigation; Behavioral: Standard of care engagement practices

INTERVENTIONS:
Behavioral: Family-based mental health navigation — Family-based navigator intervention combined with mHealth practices to improve mental health treatment initiation and engagement
Behavioral: Standard of care engagement practices — Standard of care engagement practices and services-as-usual
  Arms: Standard of care, then family-based mental health navigation

SUMMARY:
This study will focus on developing and testing a family-based mental health navigator intervention, the Foster Care Family Navigator (FCFN), to evaluate whether the intervention combined with mHealth would be efficacious in improving mental health service initiation and engagement for child welfare-involved youth.

DETAILED DESCRIPTION:
The study will demonstrate how a family-based navigator intervention combined with mHealth may lead to improved mental health treatment initiation and engagement among child welfare-involved (CWI) youth. CWI youth have high rates of mental health symptoms relative to youth in the community, and are disproportionately racial and ethnic minorities, only perpetuating disparities in this population's mental health access and engagement. The proposed project will develop and test a family-based navigator intervention, the Foster Care Family Navigator (FCFN), a natural fit for improving CWI youth mental health service and clinical outcomes. The study will start with identifying the feasibility and acceptability of the FCFN intervention. Then, the study will determine whether the FCFN intervention improves CWI youth mental health treatment initiation and engagement, relative to standard of care (not participating in FCFN intervention). Finally, the study will characterize patterns of pre- and post-service outcomes along the behavioral health services cascade of care, to further evaluate the feasibility, acceptability, and preliminary impact of the FCFN model.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking youth
* Ages 12-17
* Have an active dependency petition with the SF Unified Family Court (newly filed or existing when the trial starts)
* Are open to SF DPH Foster Care Mental Health Clinic services
* Have an involved caregiver/legal guardian for consent
* Family has mobile phone access

Exclusion Criteria:

* Youth is not English-speaking
* Caregiver has impairment that would preclude providing informed consent
* Unavailable guardian for consent

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 124 (Actual)
Dates: Start 2020-08-20 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Time to treatment referral | 12 months post enrollment
  Number of days until treatment referral is made
Time to treatment initiation | 12 months post enrollment
  Number of days until attendance at first treatment session
Treatment engagement | 12 months post enrollment
  Engagement as measured by attendance in treatment for 6 or more weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marina Tolou-Shams, Ph.D, Principal Investigator — UC San Francisco
Locations (1):
- UCSF Zuckerberg San Francisco General Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tolou-Shams M, Ramaiya M, Lara Salas J, Ezimora I, Shumway M, Duerr Berrick J, Aguilera A, Borsari B, Dauria E, Friedling N, Holmes C, Grandi A. A Family-Based Mental Health Navigator Intervention for Youth in the Child Welfare System: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2023 Sep 12;12:e49999. doi: 10.2196/49999. PMID 37698896